CLINICAL TRIAL: NCT02864303
Title: Predictive Value of the Aβ Peptides Salivary Dosage for Alzheimer's Disease Diagnosis
Brief Title: Use of Saliva for Alzheimer's Disease Diagnosis
Acronym: SalivALZ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of the inclusion period
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8835
Record Dates: First submitted 2016-07-27; First posted 2016-08-12 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Mild Cognitive Impairment; Saliva; Amyloid peptides; Diagnosis
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Alzheimer disease (Other): Saliva samples were collected on this patients
  Interventions: Other: Saliva samples

INTERVENTIONS:
Other: Saliva samples — saliva specimens were collected using a neutral or citric acid impregnated Salivette cotton swabs on Alzheimer patients to quantify the level of amyloid peptides

SUMMARY:
Although saliva is not generally regarded as one of the most interesting biological fluids, the fact that it can be sampled using simple, noninvasive methods makes it an interesting alternative to cerebrospinal fluid (CSF) or blood for diagnostic purposes. The use of salivary diagnostics is moreover increasing these past 10 years, as shown with the abundant literature as well as various clinical trials. Saliva collection which is now well standardized has the major advantage of being simple and non-invasive. An original study had already discussed possible changes in the salivary composition in Alzheimer's disease (AD). The feasibility and the potential interest of measuring saliva concentration of the amyloid peptides was reported in an article published recently. The prospect of using saliva for early diagnosis and monitoring of AD is thus of major interest and the objective of the current trial.

DETAILED DESCRIPTION:
Saliva samples

To minimize the circadian effects, saliva specimens were all collected between 9:00 and 11:00 a.m. Prior to the sampling procedure, participants rinsed out their mouths three times with water. To induce salivary production, patients were asked to chew neutral or citric acid impregnated Salivette cotton swabs for exactly 60 seconds. Saliva specimens were centrifuged for 2 minutes at a rate of 1000 g to yield clear saliva, which was aliquoted into 500 µL samples in LoBind tubes and stored at -80°C before being analyzed.

Design of the study

Saliva sampling will be performed at V0 (M0), V1 (M12) and V2 (M24). Blood sampling will take place also in V1 (M12). The cases and the controls will be systematically reviewed 12 months after inclusion with a new saliva collection and a cognitive assessment (for cases and controls).

Amyloid peptide quantification

Levels of human endogenous Aβ40 and Aβ42 in saliva and human plasma samples are determined with human specific enzyme-linked immunosorbent assay (ELISA) (Biosource International, Invitrogen), according to the manufacturer's instructions. Briefly, 50 μl of saliva and plasma samples were added in triplicate to the microtiter wells. Detection limit of the assay was 6 pg/ml for Aβ40 and 1 pg/ml for Aβ42.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women;
* Aged ≥ 55 years and 80 years;
* Patients mild cognitive impairment (MCI), not answering either the criteria of a normal cognitive functioning or the criteria of the insanity, but meeting the criteria of diagnosis of following MCI in the term of a complete cognitive balance sheet (assessment) and according to the diagnostic procedure published by the work group on the MCI of the EADC:

  * Mnesic complaint
  * Decline of the cognitive performances with regard to the previous capacities
  * Cognitive disorders(confusions) objectified by the clinical evaluation (change of the memory and/or another cognitive sphere)
  * The cognitive change has no echo on the everyday life
  * Not dementia syndrome
* Signature of the informed consent by the patient;
* Subject affiliated to a national insurance scheme.

Exclusion Criteria:

* Edentulous total or poor oral hygiene;
* Absence of the signed informed consent;
* Clinical and laboratory information insufficient or unavailable;
* Patient deprived of freedom, by court or administrative order;
* Major protected by law;
* Presence of a contagious viral affection (HIV, hepatitis B and C);
* Patient included in a therapeutic trial targeting the metabolism of metabolism of amyloid peptides ;
* Patient in period of relative exclusion with regard to another protocol or for which the annual maximum amount of the 4500-compensations was reached.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Aβ40 and Aβ42 | 24 months
  Amyloid quantification using ultra sensitive immunoassays

SECONDARY OUTCOMES:
Neuropsychologic tests | 24 months
  Neuropsychologic questionaries assessed on the Alzheimer patients
ApoE polymorphism | 24 months
  Measure of the ApoE polymorphism by biological analyses

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Lehmann, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHRU, Montpellier, France

IPD SHARING:
Plan to Share IPD: No